CLINICAL TRIAL: NCT02001415
Title: Randomized Controlled Trial of Different Lens Treatments on Chinese Adolescent Myopia
Brief Title: Efficacy Study of Different Lens Treatments on Chinese Adolescent Myopia
Acronym: DLTCAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Z131107002213127
Record Dates: First submitted 2013-11-23; First posted 2013-12-04 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Progressive Myopia
Keywords: Progressive Myopia; Contact Lenses; Spectacles
MeSH Terms: conditions — Myopia, Degenerative | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Spectacles (Active Comparator): Spectacles are the most common lens treatment to correct myopia. This arm is set to be as a control group for the other two arms. Myopia patients who enter in this group will wear a normal pair of glasses after the baseline examinations (axial length, refraction...).
  Interventions: Other: Spectacles
- Myovison (Active Comparator): Myovision is a kind of specially designed, commercially available spectacle lenses that could control the peripheral refraction of myopia patients. Latest studies have changed the understanding of myopia--correcting both central and peripheral vision during lens treatment is indicating to be an effective way of slowing down eye growth. Patients who entered this group will wear a pair of Myovision after baseline examinations.
  Interventions: Other: Myovision
- Ortho-K (Active Comparator): Orthokeratology has recently been reported as an effective way to control eye growth for myopia adolescents. Patents who enter this group will wear ortho-K lenses during sleep after baseline examinations.
  Interventions: Other: Orthokeratology

INTERVENTIONS:
Other: Spectacles — Normal spectacle lenses were used to correct myopia as the control group.
  Arms: Spectacles
Other: Myovision — Myovision is a kind of specially designed spectacle glasses that could control the peripheral refraction of myopia patients. It is commercially available.
  Arms: Myovison
Other: Orthokeratology — Orthokeratology lenses.
  Arms: Ortho-K

SUMMARY:
The purpose of this study is to determine the efficacy of different lens treatments (normal spectacle lens, ortho-K, & Myovision) on myopia control in Chinese adolescent patients.

DETAILED DESCRIPTION:
Different lens treatments include normal spectacle lens, orthokeratology, and Myovision (a specially designed spectacle lens commercially available with peripheral defocus controlled as relative myopia).

This study is to evaluate the efficacy of these three methods in controlling myopia progression. Until now, there is no sufficient clinical evidences to compare different lens treatments.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent myopia patients
* Myopic refraction between -1.00D and -4.50D
* Astigmatism equal or less than -1.50D
* Normal break up time of tear film (BUT > 10s)

Exclusion Criteria:

* Existence of any ocular diseases except ametropia
* Hyperopia
* Severe dry eye

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Change of Ocular Axial Length | Baseline, 6 months, 12 months
  Ocular axial length (AL), which increases with age, will be measured 3 times by an IOLMaster. The first AL examination was considered as the baseline data, and will be repeated 6 and 12 months later.

SECONDARY OUTCOMES:
Change of Spherical Equivalent Refraction | Baseline, 6 months, 12 months
  Spherical Equivalent Refraction (SER), which usually changes from time to time, will be measured 3 times by an open field auto-refractometer. The first SER examination was considered as the baseline data, and will be repeated 6 and 12 months later.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Wang, Dr., Principal Investigator — Peking University People's Hospital
Locations (1):
- Ophthalmology Department of Peking University People's Hospital, Beijing, China